CLINICAL TRIAL: NCT06571968
Title: Accuracy of Computer Guided Four Implants Placement in Completely Edentulous Mandible by Using Fully Versus Semi Guided Prototyped Surgical Stent
Brief Title: Accuracy of Computer Guided Four Implants Placement in Completely Edentulous Mandible
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: M05010322
Record Dates: First submitted 2024-08-08; First posted 2024-08-26 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2024-07

CONDITIONS: Implant Placement
Keywords: Fully-guided surgical stent; semi-guided surgical stent; accuracy analysis

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical trial
Who Masked: Investigator
Masking Description: Dental professionals who were not informed about the group assignments carried out the assignment and randomization of patients to the treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- fully guided surgical technique (Other): The guides were designed with metal sleeves for guided drilling and guided implant placement and additional guide sleeves for the stabilization of the template by fixation screws.The implant width and length were selected for each patient according to previous 3d cone beam, and the drills of this kit were 11 mm longer than conventional drills. The surgery was performed without flap elevation. The guide was seated and fixed by means of 2-mm cortical screws in the buccal region after using of the corresponding drills.
  Interventions: Device: fully guided stent
- semi guided surgical technique (Other): The guides were designed with metal sleeves for guided drilling and guided implant placement and additional guide sleeves for the stabilization of the template by fixation screws.The implant width and length were selected for each patient according to previous 3d cone beam, and the drills of this kit were 11 mm longer than conventional drills.The surgery was performed without flap elevation. The stent was removed before the final drilling
  Interventions: Device: semiguided stent

INTERVENTIONS:
Device: fully guided stent — All surgical procedures with drills were done through the stent., the implant was picked up from the implant holder and then installed, still with the surgical guide in situ, by using the ratchet and ratchet connector at a motor speed of 20 rpm, followed by cover screw placement without the need for sutures.
  Arms: fully guided surgical technique
Device: semiguided stent — The first osteotomy was performed with the surgical guide in situ using a 1.95 mm pilot-drill. Successive color coded implant drills were used to prepare implant osteotomies. When using each twist drill, a removable sleeve having a diameter to coincide with the drill and inserted into the sleeve of the surgical guide.
  The stereo lithographic guide template was removed and the receptor sites were irrigated with saline solution then the final drill of the implant system 3.5 mm diameter was used to finalize the osteotomy. The implant was gripped with the placement aid, released from the implant holder by 1/4 turn and manually inserted into the prepared implant site using a finger placement tool or hand ratchet. A torque of 45 N cm should not be exceeded during insertion procedure and cover screws were screwed over it.
  Arms: semi guided surgical technique

SUMMARY:
Thirty-six completely edentulous healthy patients received four mandibular implants and were randomly divided into the following groups: (A) The implants were installed by fully guided stereolithographic stent (n = 18), and (B) The implants were installed by semi-guided stereolithographic stent. (n = 18). The accuracy analysis was performed by one experienced process engineer (DB). Cone beam computed tomography was performed before and after the surgical procedure to plan the virtual implant position and fabricate the surgical guide, as well as to determine implant position deviations. Both CBCT scans were superimposed, and the software compared preoperative linear and angular virtual measurements of planned implants with real measurements of the placed implants.

DETAILED DESCRIPTION:
Objectives: Current study aimed to assess the accuracy of fully- guided implant placement in completely lower edentulous patients compared to the semi-guided protocol.

Materials and Methods: Thirty-six completely edentulous healthy patients received four mandibular implants and were randomly divided into the following groups: (A) The implants were installed by fully guided stereolithographic stent (n = 18), and (B) The implants were installed by semi-guided stereolithographic stent. (n = 18). The accuracy analysis was performed by one experienced process engineer (DB). Cone beam computed tomography was performed before and after the surgical procedure to plan the virtual implant position and fabricate the surgical guide, as well as to determine implant position deviations. Both CBCT scans were superimposed, and the software compared preoperative linear and angular virtual measurements of planned implants with real measurements of the placed implants. Measurements and analysis of results were performed by means of a software tool used during virtual planning (P3Dental; Protótipos).

ELIGIBILITY:
inclusion criteria:

* All patient wearing maxillary conventional denture.
* All patients had temporary mandibular overdenture supported by vertically inserted 4-implant at least six months ago.
* They were healthy, free from any systemic diseases relating to bone resorption such as uncontrolled diabetics or osteoporosis. This was achieved through medical history and clinical examination by physician.
* All patients are of angel's class I maxillo-mandibular relationships.

Exclusion Criteria:

* Patients had head and neck radiotherapy, patients with bleeding disorders or hepatic patients.
* Patients with metabolic disorders as diabetes mellitus, osteoporosis and hepatic disorders that might affect osseointegration.
* Long term immunosuppress and corticosteroid drug therapy.
* Patient with abnormal habits as clenching and bruxism.
* Smoking patient.
* Patient with problems in TMJ

Ages: 58 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-05-14 (Actual); Primary Completion 2024-01-03 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Radio graphic evaluation (Angular deviation) | one year
  For both groups, postoperative CBCT scan was performed after implant placement. The same parameters of preoperative CBCT were followed according to the patient's position, image acquisition, and use of the same apparatus. This scan was performed with the same dental prosthesis as that used for the initial preoperative CBCT scanning, equipped with the gutta percha references, for superimposition of the images. The previously fabricated occlusal registration was used to align the prosthesis. Both CBCT scans were superimposed, and the software compared preoperative horizontal (Mesiodistal and buccolingual), vertical and angular virtual measurements of planned implants with real measurements of the placed implants.

SECONDARY OUTCOMES:
Radio graphic evaluation (linear deviation) | one year
  For both groups, postoperative CBCT scan was performed after implant placement. The same parameters of preoperative CBCT were followed according to the patient's position, image acquisition, and use of the same apparatus. This scan was performed with the same dental prosthesis as that used for the initial preoperative CBCT scanning, equipped with the gutta percha references, for superimposition of the images. The previously fabricated occlusal registration was used to align the prosthesis. Both CBCT scans were superimposed, and the software compared preoperative horizontal (Mesiodistal and buccolingual) measurements of planned implants with real measurements of the placed implants.

CONTACTS AND LOCATIONS:
Overall Officials: marwa aboelez, Phd, Study Chair — Mansoura University; Hassan Kheriba, Msd, Study Director — Mansoura University
Locations (1):
- Marwa Aboelez, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
statistical analysis plan
Supporting Information: SAP
Time Frame: when summary data are published
Access Criteria: raw data , statistical tests

REFERENCES:
- [Background] Malpartida-Carrillo V, Tinedo-Lopez PL, Ortiz-Culca F, Guerrero ME, Amaya-Pajares SP. Techniques for retrievability and for registering screw access holes in cement-retained implant-supported prostheses: A scoping review of the literature. J Prosthet Dent. 2020 Mar;123(3):427-433. doi: 10.1016/j.prosdent.2019.03.011. Epub 2019 Jul 12. PMID 31307803